CLINICAL TRIAL: NCT03262142
Title: Targeted AntiBiotics for Chronic Pulmonary Disease: Can Targeted Antibiotic Therapy Improve the Prognosis of Pseudomonas Aeruginosa Infected Patients With Chronic Pulmonary Obstructive Disease, Non-cystic Fibrosis Bronchiectasis and Asthma? A Multicenter, Randomized, Controlled, Open-label Trial.
Brief Title: Targeted AntiBiotics for Chronic Pulmonary Diseases
Acronym: Target-ABC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Josefin Eklöf, Principal Investigator, Chronic Obstructive Pulmonary Disease Trial Network, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: coptrin2
Record Dates: First submitted 2017-08-21; First posted 2017-08-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: COPD; Respiratory Tract Infections; Pseudomonas Aeruginosa; Bronchiectasis; Asthma
Keywords: chronic pulmonary disease; Pseudomonas Aeruginosa
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Tract Infections; Pseudomonas Infections; Bronchiectasis; Asthma | interventions — Piperacillin, Tazobactam Drug Combination; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard antibiotic treatment (Active Comparator): Intravenous Piperacillin/tazobactam + oral Ciprofloxacin for 14 days
  Interventions: Drug: Piperacillin/tazobactam; Drug: Ciprofloxacin
- Antibiotic-free treatment (No Intervention): No antibiotic treatment

INTERVENTIONS:
Drug: Piperacillin/tazobactam — Intravenous Piperacillin/tazobactam four times daily
  Arms: Standard antibiotic treatment
Drug: Ciprofloxacin — Oral Ciprofloxacin twice daily
  Arms: Standard antibiotic treatment

SUMMARY:
This is a prospective, randomized multi-center trial investigating the impact of lower airway infection with P. aeruginosa in COPD patients. The aim of the study is to evaluate if targeted antibiotic therapy against P. aeruginosa can improve the prognosis in patients with COPD. non-CF bronchiectasis (BE) and asthma.

DETAILED DESCRIPTION:
P. aeruginosa represents a potentially significant cause of acute exacerbation of chronic pulmonary diseases and is possibly associated with significant morbidity and mortality. Despite this, the role of P. aeruginosa in the course of COPD, non-CF BE and asthma is less well characterized, and evidence based guidelines for management and treatment of the bacteria are lacking.

P. aeruginosa is more likely to be isolated from patients with more advanced disease and severely impaired lung function. It is, however, difficult to draw definitive conclusions regarding the extent to which the bacteria contributes to adverse clinical outcomes since severely reduced lung function by itself is a strong predictor of mortality in patients with chronic pulmonary disease. Infection with P. aeruginosa might therefore be secondary to damaged lung tissue and decreased lung function, and thereby have no independent impact on the prognosis

So far, and to the investigators best knowledge, no randomized controlled trial has been conducted to investigate whether specific antibiotic treatment of P. aeruginosa can reduce the risk of new exacerbations and improve the long-term prognosis in patients with COPD, non-CF BE and asthma.

In Denmark, the first choice of treatment for P. aeruginosa is usually a 10-14 day therapy of intravenous combination treatment of P. aeruginosa active antibiotics (piperacillin/tazobactam and ciprofloxacin).

The aim of the study is to investigate whether the intervention with targeted pseudomonas active antibiotics can reduce the loss of lung function, reduce the frequency of exacerbations and mortality.

ELIGIBILITY:
Inclusion Criteria:

* P. aeruginosa-positive lower respiratory tract sample.
* COPD, non-CF bronchiectasis, or asthma verified by a respiratory specialist based on clinical assessment and additional tests: COPD: spirometry; Asthma: reversibility; Non-CF bronchiectasis: high-resolution computed tomography scan.
* Minimum of two previous exacerbations, or one previous hospitalization-requiring or emergency room-demanding exacerbation, with the treatment of systemic prednisolone and/or antibiotics within the last 12 months.
* Written informed consent

Exclusion Criteria:

* Immune-modulating therapy (except ≤ 10 mg prednisolone/day)
* Men < 40 years
* Women <= 55 years
* Non- menopausal women > 55 years
* Life expectancy < 90 days
* Severe mental illness
* Severe language difficulties or inability to provide informed consent
* Known drug allergy to 1) Fluoroquinolones and 2) both Piperacillin/tazobactam, Cephalosporins and Carbapenems
* Attempted eradication of P. aeruginosa x 2 within the last 12months, or completed eradication therapy within the last 14 days
* The investigator 's opinion is that the participant requires antibiotic treatment. This exclusion criterion must be discussed with the coordinating investigator before the final decision on exclusion is taken.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Time to prednisolone and/or antibiotic requiring exacerbation or death, in primary or secondary health care sectors from day 20 to day 365 from randomization. | day 20-365
  Time alive and without exacerbation between day 20-365 from the date of recruitment.
Days alive and without hospitalisation from day 20 to day 365 from randomization. | day 20-365
  Days alive and out of hospital between day 20-365 from the date of recruitment.

SECONDARY OUTCOMES:
Number of re-admissions with pulmonary exacerbation within 365 days from randomization. | 365 days
  Number of re-admissions with pulmonary exacerbation within 365 days from randomization.
Death within 365 days from randomization. | 365 days
  Death within 365 days from randomization.
Microbiological cure | 90 days
  Microbiological cure = P. aeruginosa-negative sputum culture until day 90.
  Non-microbiological cure = positive sputum culture with same P.aeruginosa clone as baseline clone ≤ day 90.
  Re-infection = positive sputum culture with different P. aeruginosa clone compare to baseline clone ≤ day 90.
Clinical cure | 14 days
  Resolution or improvement of clinical symptoms related to P. aeruginosa within day 14.
  Clinical failure = persistent of worsened clinical symptoms related to P. aeruginosa within day 14.
Number of days with non-invasive ventilation or invasive ventilation within 90 days from randomization. | 90 days
  Number of days with non-invasive ventilation or invasive ventilation within 90 days from randomization.
Change in forced expiratory volume in the first second (FEV1) from randomization to day 90. | 90 days
  Change in forced expiratory volume in the first second (FEV1) from randomization to day 90.
Decrease of ≥ 200 ml in FEV1 from randomization to day 365. | 365 days
  Decrease of ≥ 200 ml in FEV1 from randomization to day 365.
Change in COPD Assessment Test (CAT) from randomization to day 90. | 90 days
  Change in COPD Assessment Test (CAT) from randomization to day 90.
Change in body mass index (BMI) from randomization to day 90. | 90 days
  Change in body mass index (BMI) from randomization to day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik Jensen, MD, Consultant, Phd, Study Director — Chronic Obstructive Pulmonary Disease Trial Network, Denmark
Locations (1):
- Herlev and Gentofte Hospital, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Eklof J, Alispahic IA, Sivapalan P, Wilcke T, Seersholm N, Armbruster K, Kjaergaard JL, Saeed MI, Nielsen TL, Browatzki A, Overgaard RH, Fenlev CS, Harboe ZB, Andreassen HF, Lapperre TS, Pedersen L, Johnsen S, Ulrik CS, Janner J, Moberg M, Heidemann M, Weinreich UM, Vijdea R, Linde H, Titlestad I, Johansson SL, Rosenvinge FS, Ostergaard C, Ghathian KSA, Gundersen L, Christensen CW, Bangsborg J, Jensen TT, Sorensen VM, Ellingsgaard T, Datcu R, Coia JE, Bodtger U, Jensen JUS. Targeted AntiBiotics for Chronic pulmonary diseases (TARGET ABC): can targeted antibiotic therapy improve the prognosis of Pseudomonas aeruginosa-infected patients with chronic pulmonary obstructive disease, non-cystic fibrosis bronchiectasis, and asthma? A multicenter, randomized, controlled, open-label trial. Trials. 2022 Sep 27;23(1):817. doi: 10.1186/s13063-022-06720-z. PMID 36167555
- [Derived] Eklof J, Alispahic IA, Armbruster K, Lapperre TS, Browatzki A, Overgaard RH, Harboe ZB, Janner J, Moberg M, Ulrik CS, Andreassen HF, Weinreich UM, Kjaergaard JL, Villadsen J, Fenlev CS, Jensen TT, Christensen CW, Bangsborg J, Ostergaard C, Ghathian KSA, Jordan A, Klausen TW, Nielsen TL, Wilcke T, Seersholm N, Sivapalan P, Jensen JS. Systemic antibiotics for Pseudomonas aeruginosa infection in outpatients with non-hospitalised exacerbations of pre-existing lung diseases: a randomised clinical trial. Respir Res. 2024 Jun 6;25(1):236. doi: 10.1186/s12931-024-02860-9. PMID 38844921
- [Derived] Eklof J, Misiakou MA, Sivapalan P, Armbruster K, Browatzki A, Nielsen TL, Lapperre TS, Andreassen HF, Janner J, Ulrik CS, Gabrielaite M, Johansen HK, Jensen A, Nielsen TV, Hertz FB, Ghathian K, Calum H, Wilcke T, Seersholm N, Jensen JS, Marvig RL. Persistence and genetic adaptation of Pseudomonas aeruginosa in patients with chronic obstructive pulmonary disease. Clin Microbiol Infect. 2022 Jul;28(7):990-995. doi: 10.1016/j.cmi.2022.01.017. Epub 2022 Feb 3. PMID 35124256
- [Derived] Eklof J, Sorensen R, Ingebrigtsen TS, Sivapalan P, Achir I, Boel JB, Bangsborg J, Ostergaard C, Dessau RB, Jensen US, Browatzki A, Lapperre TS, Janner J, Weinreich UM, Armbruster K, Wilcke T, Seersholm N, Jensen JUS. Pseudomonas aeruginosa and risk of death and exacerbations in patients with chronic obstructive pulmonary disease: an observational cohort study of 22 053 patients. Clin Microbiol Infect. 2020 Feb;26(2):227-234. doi: 10.1016/j.cmi.2019.06.011. Epub 2019 Jun 22. PMID 31238116
- See also: Related Info — http://coptrin.dk/